CLINICAL TRIAL: NCT05394558
Title: A Phase Ib/II Study on AsiDNA in Association With Re-irradiation in Children, Adolescents and Young Adults With High-grade Glioma
Brief Title: AsiDNA Children, Adolescents and Young Adults
Acronym: AsiDNA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IDMC recommendations
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IC 2020-21
Record Dates: First submitted 2021-12-16; First posted 2022-05-27 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Recurrent High-grade Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy + AsiDNA (Experimental): Patients will receive the IMP which is the AsiDNA (etidaligide). AsiDNA will be administered intravenously as a 1-hour infusion. All patients will receive a loading dose for three consecutive days, with Day 1 being the start day of radiotherapy, followed by once weekly administrations during 11 weeks.
  The infusion of AsiDNA should be administered between 4 and 6 hours before the planned start of radiotherapy.
  After the administration of AsiDNA, Patients with DIBG will receive a total dose of 18 Gy, delivered in 10 fractions of 1.8 Gy, i.e. 5 fractions per week for 2 weeks, starting on Day 1. Patients with supratentorial non-DMG or DMG will receive a total dose of 36 Gy, delivered in 20 fractions of 1.8 Gy, i.e. 5 fractions per week for 4 weeks, starting on Day 1.
  Interventions: Drug: AsiDNA
- Radiotherapy (Active Comparator): Patients with DIBG will receive a total dose of 18 Gy, delivered in 10 fractions of 1.8 Gy, i.e. 5 fractions per week for 2 weeks, starting on Day 1. Patients with supratentorial non-DMG or DMG will receive a total dose of 36 Gy, delivered in 20 fractions of 1.8 Gy, i.e. 5 fractions per week for 4 weeks, starting on Day 1.
  Interventions: Drug: AsiDNA

INTERVENTIONS:
Drug: AsiDNA — Administration of AsiDNA followed by radiotherapy

SUMMARY:
HGG comprises diffuse midline gliomas (DMG), including diffuse infiltrating brainstem glioma (DIPG), characterised by histone gene mutations, as well as non-DM HGGs mainly in non-midline supratentorial areas, with distinct molecular abnormalities. First-line treatment comprises surgery when doable (non-DM HGGs), and radiotherapy in all cases. Chemotherapy or other drugs in clinical trials may be added during and/or after radiotherapy depending on the HGG subtype. The recurrence rate is nevertheless high in all paediatric and adolescent HGGs. If the time interval between the end of first-line radiotherapy and relapse is long enough, re-irradiation often provides good palliation of symptoms, delays disease progression, improves quality of life and has minimal and manageable toxicity. Nevertheless, strategies to increase efficacy without increasing toxicity in the treatment of recurrent paediatric HGG are much needed.

AsiDNA™ is a DNA repair inhibitor that increases the vulnerability of tumour cells to irradiation without increasing toxicity in healthy tissues. Its novel mechanism of action, based on perturbation of the DNA damage recognition steps in DNA repair, makes its activity specific to tumour cells. Intravenous administration of AsiDNA is currently being investigated in adults with advanced solid tumours. The MTD was not reached during the escalating dose study on the safety, pharmacokinetics and pharmacodynamics of AsiDNA administered as a 1-hour infusion, however an optimal dose range (400-600 mg) was identified for further development, based on the favourable safety and PK profiles. Preclinical studies on AsiDNA added to radiotherapy have shown increased survival and no increase in short- or long-term toxicity due to the high doses of irradiation.

The study will provide paediatric patients who have recurrent HGG with early access to innovation, even during the early drug development stage in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from patient (depending on age) and/or parents or legal guardian;
2. Patient must be ≥ 12 months and < 25 years of age at the time of enrolment on the study;
3. Recurrent high-grade glioma (HGG), including diffuse midline glioma (DMG) and non-DMG, based on RAPNO criteria confirmed by central radiological review, with or without histology if biopsy performed prior to inclusion;
4. Available tumour material, at least paraffin embedded and/or also frozen material;
5. For DMG and non-DMG HGG, prior radiation dose prescribed ≤ 60 Gy, completed at least 6 months prior to inclusion, with stable disease;
6. Maximum cumulative radiation dose to optic chiasm and optic nerve < 56 Gy and < 54 Gy to upper cervical spine (at level C1);
7. Life expectancy > 2 months at Screening;
8. Patient must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of ≥ 50 % , not taking into account neurological deficit;
9. No significant abnormality on laboratory tests at Screening, including:

   1. Haemoglobin > 9 g/dL;
   2. Neutrophils > 1.0 x 109/L;
   3. Platelets > 100 x 109/L;
   4. Total bilirubin < 1.5 x ULN;
   5. AST and ALT< 2.5 x ULN;
   6. Serum creatinine < 1.5 x ULN for age;
   7. Normal coagulation tests.
10. No organ toxicity > grade 2 according to NCI CTCAE version 5.0 classification, notably cardiovascular, pulmonary or renal diseases, including congenital QT prolongation syndrome, nephrotic syndrome, glomerulopathy, uncontrolled high blood pressure despite appropriate treatment, interstitial pulmonary disease, pulmonary hypertension;
11. Negative serum pregnancy test for women of child-bearing potential, and highly effective birth control method for male and female patients of reproductive potential;
12. Patients covered by social security or health insurance in compliance with the national legislation relating to biomedical research.

Exclusion Criteria:

5. Prior radiation dose prescribed > 60 Gy; 6. Massive intra-tumour haemorrhage; 7. Pseudoprogression (including after central review); 8. Metastatic relapse; 9. Other anticancer treatment, on-going or within less than 4 weeks prior to inclusion; 10. Prior or concurrent malignant disease, other than HGG, diagnosed or treated within 5 years prior to inclusion; patients with CMMRD are eligible; 11. Uncontrolled intercurrent disease or active infection; 12. Concomitant disease or other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study; 13. Patients unable to comply with the protocol for any reason; 14. Organ toxicity > grade 2 according to NCI CTCAE version 5.0 classification, notably cardiovascular, pulmonary or renal diseases, including congenital QT prolongation syndrome, nephrotic syndrome, glomerulopathy, uncontrolled high blood pressure despite appropriate treatment, interstitial pulmonary disease, pulmonary hypertension 15. Breastfeeding or pregnancy

Ages: 12 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
DLT(Dose-Limiting Toxicities) | 8 weeks after treatment initiation
  Dose-limiting toxicities, i.e. grade ≥ 3 toxicities according to NCI-CTCAE version 5.0, considered as at least possibly related to the treatment during the 8 weeks after treatment initiation.
Activity | 3 months after treatment initiation
  3-month progression-free survival (PFS), i.e. the probability for a patient to be alive and free of disease progression based on clinical or radiological criteria, or death from any cause at 3 months after inclusion in the study. Radiological progression will be assessed using RAPNOHGG criteria. Patients lost to follow-up will be counted as failures at the last assessment date.

SECONDARY OUTCOMES:
Late Onset toxicity | 8 weeks and until 12 months after treatment initiation
  Late-onset toxicity, defined as any toxicity, i.e. any AE considered as at least possibly related to treatment, that occurs more than 8 weeks after treatment initiation;
MR pattern of disease response and of potential treatment-related toxicity, | 3 months after treatment initiation
  MR pattern of disease response and of potential treatment-related toxicity, assessed by central review based on morphological and functional imaging features present on the various MR examinations;
Best objective Response Rate | 3 months after treatment initiation
  Best objective response rate, defined as the percentage of patients with complete or partial responses according to RAPNO criteria as assessed by the investigator
Overall survival | 12 months after treatment initiation
  Overall survival, defined as the time from inclusion in the study to death from any cause.
  Patients alive or lost to follow-up at the cut-off date will be censored at the last date they were known to be alive;
Palliation of symptoms 1 | 3 months after treatment initiation
  Palliation of symptoms, assessed using the Lansky Play Scale (LPS) or Karnofsky score of ≥ 50 %
Palliation of symptoms 2 | 3 months after treatment initiation
  Performance Status (KPS)
Palliation of symptoms 2 | 3 months after treatment initiation
  Need for corticosteroids and/or bevacizumab
Pharmacokinetic parameters of AsiDNA. | 1 week after treatment initiation
  Maximal observed drug concentration (Cmax);
Pharmacokinetic parameters of AsiDNA. | 1 week after treatment initiation
  absorption and elimination half-life (t1/2))
Pharmacokinetic parameters of AsiDNA. | 1 week after treatment initiation
  time to reach maximum observed drug concentration (Tmax);
Pharmacokinetic parameters of AsiDNA. | 1 week after treatment initiation
  area under the curve (AUC0-t (experimental time points)
Pharmacokinetic parameters of AsiDNA. | 1 week after treatment initiation
  AUC0-∞ (extrapolated to infinity)

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Chu Angers, Angers
  - Chru Bordeaux, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Chu La Timone Hopital Enfants, Marseille
  - Chu Nancy, Nancy
  - Institut Curie, Paris
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).